CLINICAL TRIAL: NCT05779007
Title: Assessment of the Dose Reduction and Discontinuation Associated With Anti-Fibrotic Medications in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Dose Reduction and Discontinuation With Anti-Fibrotic Medications
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0526
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone; nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pirfenidone initiators cohort: IPF patients from the Optum Research Database (ORD) who presented at least one pirfenidone prescription during the identification period (the date of first prescription for pirfenidone was considered the index date, between October 2014 up to December 2021) and with at least 12 months of continuous enrollment in the health plan during pre-and post-index period.
  Interventions: Drug: Pirfenidone
- Nintedanib initiators cohort: IPF patients from the Optum Research Database (ORD) who presented at least one nintedanib prescription during the identification period (the date of first prescription for nintedanib was considered the index date, between October 2014 up to December 2021) and with at least 12 months of continuous enrollment in the health plan during pre-and post-index period.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone
  Groups: Pirfenidone initiators cohort
Drug: Nintedanib — Nintedanib
  Groups: Nintedanib initiators cohort

SUMMARY:
The overarching aim of our study is to assess the incidence of dose reduction and discontinuations for pirfenidone and nintedanib.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one pirfenidone or nintedanib prescription during the identification period (0/01/2014 to 09/30/2021; the date of first prescription for pirfenidone/nintedanib is the index date)
* Evidence of IPF: patient with at least one inpatient or two outpatient claims (>14 days apart) with a diagnosis code for IPF during the study period (10/01/2013 to 09/30/2022)
* At least 18 years old at the index date
* Have at least 12 months of continuous enrollment in the health plan during pre-index period, and at least 6 months of continuous enrollment in post-index period

Exclusion Criteria:

* Any history of lung transplant during the 12-months pre-index/baseline period
* Any claims for a skilled nursing facility, a long-term care facility or hospice care during the 12-month pre-index period
* Evidence of non-IPF chronic fibrosis Interstitial Lung Disease (ILD) or connective tissue diseases during the 12-months pre-index period. The following conditions will be excluded: autoimmune, or connective tissue diseases (i.e., rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), dermatopolymyositis, systemic sclerosis, Sjogren's syndrome, and mixed connective tissue disease (CTD), sarcoidosis, and hypersensitivity pneumonitis).
* Missing demographic information (i.e., age or sex)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic pulmonary fibrosis (IPF) who initiated either pirfenidone or nintedanib between October 2014 and September 2021.
Sampling Method: Non-Probability Sample
Enrollment: 2778 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim, Ridgefield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a retrospective cohort study to assess the dose reduction/interruption and discontinuation with nintedanib and pirfenidone initiators among patients with Idiopathic Pulmonary Fibrosis (IPF) from the Optum Research Database (ORD) who initiated either pirfenidone or nintedanib between October 2014 and December 2021.
Pre-assignment Details: Patients with IPF who presented at least one pirfenidone or nintedanib prescription during the identification period and with at least 12 months of continuous enrollment in the health plan during pre- and post-index period. A total of 1,389 new users of nintedanib were matched to equal number of new pirfenidone users.
Period: Overall Study
Arm/Group | Nintedanib Initiators Cohort | Pirfenidone Initiators Cohort
Started | 4972 | 3398
Propensity Score Matched Patients | 1389 | 1389
Completed | 1455 | 1389
Not Completed | 3517 | 2009
Not completed — not meeting eligibility criteria | 3517 | 2009

BASELINE CHARACTERISTICS:
Population: Propensity score matched (PSM) cohorts of IPF patients between the nintedanib and pirfenidone initiators groups (1:1). Patients >= 18 years old and registered in Optum Research Database (ORD) between October 2014 and December 2021.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib Initiators Cohort | Pirfenidone Initiators Cohort | Total
Number analyzed (Participants) | 1389 | 1389 | 2778
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (7.6) | 73.9 (7.6) | 73.52 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 534 | 549 | 1083
  Male | 855 | 840 | 1695
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and Ethnicity were not collected from any participant. Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Reduction and/or Temporary Dose Reduction (Sub-optimal Dose) by 12 Months
Description: Number of patients with sub-optimal dose was be defined as patients with an average daily dose not following the prescribing information of nintedanib and pirfenidone for at least 90 consecutive days, corresponding to ≤ 66.67% dose strength for pirfenidone and ≤ 66.67% dose strength for nintedanib.
  Number of patients with sub-optimal dosing by month 12 is reported.
Time Frame: From individual index date up to 12 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib Initiators Cohort | Pirfenidone Initiators Cohort
Number analyzed (Participants) | 1389 | 1389
Participants | 301 | 373

2. Secondary Outcome: Time to Treatment Discontinuation
Description: Treatment discontinuation was defined as presence of ninety or more days gap in refilling a prescription of the drug (pirfenidone or nintedanib)
Time Frame: From individual index date up to 12 months.
Population: Propensity score matched (PSM) cohorts of IPF patients between the nintedanib and pirfenidone initiators groups (1:1). Patients >= 18 years old and registered in Optum Research Database (ORD) between October 2014 and December 2021. Only IPF patients with event were included in the analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nintedanib Initiators Cohort | Pirfenidone Initiators Cohort
Number analyzed (Participants) | 1389 | 1389
Days | 257.47 (130.29) | 246.56 (134.55)

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: This was an observational study and was not designed to assess adverse event; therefore safety reporting was not applicable for this study. Adverse events were not planned to be collected as defined in the study protocol. Adverse Events were not monitored/assessed.
Arm/Group | Nintedanib Initiators Cohort | Pirfenidone Initiators Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Healthcare claims data not designed for research, may not represent actual medication use.

Reasons for discontinuations/dose reduction could not be ascertained as are not captured in claims database (CDB).

Adverse events could not be evaluated as these are not reliably captured in CDB.

Due to lack of availability of laboratory data/clinical information, severity of IPF+results of laboratory tests were not observed.

ORD only covers patients with commercial insurance or Medicare Advantage plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT05779007/Prot_SAP_000.pdf